CLINICAL TRIAL: NCT05134376
Title: The Effect of Virtual Reality Glasses Watched With Music on Pain Perceived by Women During Episiotomy Repair, Vital Signs and Postpartum Comfort
Brief Title: Pain Perceived by Women During Episiotomy Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, Head of Otolaryngology, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AYDIN ADNAN MENDERES UNUVERSTY
Record Dates: First submitted 2021-09-14; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Virtual Reality; Birth
Keywords: Virtual Reality; labor; pain; episiotomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental study.
Masking Description: episiotomy application and intervention was done by midwives
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workgroup (Experimental): During the repair of the mediolateral episiotomy, the pregnant women included in the study group will be shown a video accompanying the acemaşîrân office with sterile virtual reality glasses with a view of nature.
  Interventions: Other: During Episiotomy Repair, Women Will Be Watching Virtual Reality Glasses Accompanied by Music
- Control (No Intervention): Unlike the experimental group, only video and music applications will not be applied to the pregnant women included in the control group. Other applications will be done in the same way.

INTERVENTIONS:
Other: During Episiotomy Repair, Women Will Be Watching Virtual Reality Glasses Accompanied by Music — Unlike the experimental group, only video and music application will not be applied to the pregnant women included in the control group. Other applications will be done exactly.
  Arms: Workgroup

SUMMARY:
This research was carried out to evaluate the effect of video and accompanying music played with virtual reality glasses during episiotomy repair on women's perceived pain, vital signs and postpartum comfort during episiotomy repair.

This research is a randomized controlled experimental study. The study was conducted on 84 pregnant women, 40 of whom were in the intervention group and 44 were in the control group.

The goals expected to be achieved during the research are; Reducing the perceived pain during episiotomy repair with video and accompanying music played with virtual reality glasses during episiotomy repair Video and accompanying music watched with virtual reality glasses during episiotomy repair increase postpartum comfort The positive effect of video and accompanying music on vital signs during episiotomy repair with virtual reality glasses

DETAILED DESCRIPTION:
Workgroup implementation steps Informed Voluntary Consent Form and Pregnancy Introductory Form (the first 8 questions of the pregnant introductory information - labor and episiotomy follow-up form) will be filled in by the researcher, to the pregnant women who were randomized daily to the study and control group by going to the clinic during the research. During the repair of mediolateral episiotomy, the pregnant women included in the study group will be shown the video accompanying the acemaşîrân makam with sterile virtual reality glasses with a view of nature. In the literature, it is stated that the video watched with the acemaşîrân makam and virtual reality glasses reduces pain [6, 7, 21] After the internet connection is established with a smart phone, the video to be clicked on youtube.com will be clicked, Relaxation Project 1 (SBS VR) video and Acemaşiran Ayini Şerifi Ney-Bendir will be selected for the sound, and video and music will be played with virtual reality glasses by pressing the play button[22, 23] Sound and image will be adjusted as the pregnant woman wants. During the study, all pregnant women included in the study will be given the same care and follow-up, apart from watching the video. The video containing nature scenes prepared by the researcher and the acemaşîrân maqam will be watched from the moment the episiotomy is opened to the time when the episiotomy is closed. Numerical pain assessment scale will be applied before, during (during hymen suturing) and 1 hour after the end of mediolateral episiotomy repair. Postpartum comfort scale 4-24th postpartum. The vital signs of the pregnant women in the study group will be recorded by the researcher before and during episiotomy repair (during hymen suturing) and 1 hour after the end of mediolateral episiotomy repair. In episiotomy repair, the time from the first suture to the last column will be recorded. The pregnant woman will be asked how long she perceives the duration of episiotomy.

Control group application steps Unlike the experimental group, only video and music applications will not be applied to the pregnant women included in the control group. Other applications will be made in the same way.

ELIGIBILITY:
Inclusion Criteria:

* Turkish,
* 18 - 35 years
* primiparous,
* gestational week 37- 42
* Mediolateral episiotomy performed
* pregnant women in active phase Exclusion Criteria
* high risk pregnancy
* vision and hearing problem
* with deep laceration
* 3rd and 4th degree laceration

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primipary
Enrollment: 84 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | before the episiotomy intervention,
  In the numerical evaluation scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
Numerical Pain Rating Scale | during the hymen suturing during the episiotomy,
  In the numerical evaluation scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
Numerical Pain Rating Scale | one hour after the intervention.
  In the numerical evaluation scale, pain ranges from 0 (absence of pain) to 10 (unbearable pain).
Postpartum Comfort Scale | after 24 hours
  The lowest score to be taken on the scale is 34, and the highest score is 170.
Systolic Blood Pressure | before the episiotomy intervention,
  mmHg;
diastolic Blood Pressure | before the episiotomy intervention,
  mmHg;
Systolic Blood Pressure | during the hymen suturing during the episiotomy,
  mmHg;
diastolic Blood Pressure | during the hymen suturing during the episiotomy, n
  mmHg;
Systolic Blood Pressure | one hour after the intervention
  mmHg;
diastolic Blood Pressure | one hour after the intervention
  mmHg;
pulse, | before the episiotomy intervention, during the hymen suturing during the episiotomy, and one hour after the intervention
  minute;
espiratory rate | before the episiotomy intervention,
  unit
espiratory rate | during the hymen suturing during the episiotomy,
  unit
espiratory rate | one hour after the intervention
  unit

CONTACTS AND LOCATIONS:
Overall Officials: mine gökduman keleş, 1, Study Director
Locations (1):
- Adnan Menderes University Institute of Health Sciences ile, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gokduman Keles M, Altinkaya SO. The Effect of Virtual Reality Accompanied by Music on Women's Perceived Pain, Postpartum Comfort During Episiotomy Repair: A Randomized Controlled Trial. Pain Manag Nurs. 2025 Aug;26(4):e398-e404. doi: 10.1016/j.pmn.2025.02.004. Epub 2025 Mar 12. PMID 40082095